CLINICAL TRIAL: NCT04268186
Title: Noninvasive Brain Stimulation as a Tool to Study the Role of Motivation in Age-related Cognitive Abilities
Brief Title: TDCS to Improve Motivation and Memory in Elderly (TIME)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northeastern University (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sumientra Rampersad, Research Assistant Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18-07-20; R21AG061743 (NIH)
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Motivation
Keywords: cognitive functioning; elderly; healthy; tDCS; motivation; memory; structural MRI; resting-state fMRI
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Direct tDCS (Experimental): Transcranial direct current stimulation (tDCS) was computationally optimized to target mid-cingulate cortex directly.
  Interventions: Device: Direct tDCS
- Indirect tDCS (Experimental): Transcranial direct current stimulation (tDCS) was computationally optimized to target the middle frontal gyrus, a brain area connected to mid-cingulate cortex.
  Interventions: Device: Indirect tDCS
- Personalized tDCS (Experimental): Transcranial direct current stimulation (tDCS) will be individually optimized to simultaneously stimulate key nodes connected to mid-cingulate cortex, including anterior insula, MFG and supramarginal gyrus.
  Interventions: Device: Personalized tDCS
- Sham tDCS (Sham Comparator): Placebo transcranial direct current stimulation (tDCS) will be applied.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Direct tDCS — Transcranial direct current stimulation (tDCS) will be applied. Stimulation amplitude is 2 mA. Stimulation duration is 20 minutes. The configuration used is two electrodes at AFz and CPz of the 10-10 electrode system.
  Arms: Direct tDCS
Device: Indirect tDCS — Transcranial direct current stimulation (tDCS) will be applied. Stimulation amplitude is 2 mA. Stimulation duration is 20 minutes. The configuration used is two electrodes at AF3 and AF4 of the 10-10 electrode system.
  Arms: Indirect tDCS
Device: Personalized tDCS — Transcranial direct current stimulation (tDCS) will be applied. Stimulation amplitude is 2 mA. Stimulation duration is 20 minutes. The configuration used will be optimized to stimulate key nodes connected to MCC, including anterior insula, MFG and supramarginal gyrus, and designed using an individual head model that will be combined with each subject's measured connectivity map. The number of electrodes will be minimally 2 and maximally 32.
  Arms: Personalized tDCS
Device: Sham tDCS — Transcranial direct current stimulation (tDCS) will be applied. Stimulation amplitude is 2 mA. Stimulation duration is 20 minutes. Placebo stimulation will be applied by ramping the current up and immediately down over 30 seconds. The configuration used is two electrodes at AF3 and AF4 of the 10-10 electrode system.
  Arms: Sham tDCS

SUMMARY:
Fundamental advancements in understanding successful aging are limited by the lack of causal, rather than just correlational methods to connect age-related changes in memory ability to changes in brain structure and function. In this study, non-invasive electric brain stimulation will be used as a tool to create causal links between successful memory function in aging and brain structures associated with motivation. Recently, it was shown that a group of elderly, dubbed "superagers", are indistinguishable from young adults in memory performance and the structure of cortical limbic regions. A key superaging region is mid-cingulate cortex (MCC), a brain structure associated with motivation and tenacity. The MCC is a hub region that synchronizes information flow between three core brain networks. The goal of the research is to explore the contribution of motivation to memory performance by modulating MCC connectivity with transcranial direct current stimulation (tDCS) to provide the first causal evidence that experimentally induced motivation can improve memory performance. Since MCC has not been stimulated with tDCS before, we will test three different stimulation protocols and compare against a placebo. The stimulation protocols were computationally optimized for this project. The primary aim is to find the stimulation protocol most successful at improving memory performance. In order to elucidate the mechanisms behind these changes, effects of stimulation on motivation and network connectivity will be investigated. If indeed memory can be improved by increasing motivation and effort via stimulating MCC, this study will generate new insights into the motivational mechanisms of successful aging.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 65 and 80
* normal or corrected to normal vision
* fluent in speaking, reading and understanding English
* right-handed

Exclusion Criteria:

* any metal implants that may cause harm through MRI scanning
* other metals that may interfere with obtaining MRI signals
* claustrophobic
* pregnancy
* history of neurological or psychiatric illnesses
* history of fainting, seizures or epilepsy
* history of migraines
* history of drug abuse
* learning disability
* intracranial lesion
* any prescription or regular medication except for birth control
* any uncontrolled medical condition
* skin disease or damage on scalp
* hair style or head dress that prevents electrode contact with the scalp
* any condition affecting agility of hands (e.g. acute or chronic tenosynovitis, active joint deformity of arthritic origin)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in "Feeling of difficulty" from baseline | 1 week
  Self-reports of difficulty will be queried during a memory task. Feeling of difficulty asks "How easy or difficult do you think the task will be (did you find the task)?" Answer is reported on a 7 point-scale.
Change in "Estimates of effort" from baseline | 1 week
  Self-reports of effort will be queried during a memory task. Estimates of Effort asks "How much effort do you think it will take you (did it take you) to complete the task?" Answer is reported on a 7 point-scale.
Change in "NASA Task Load Index" from baseline | 1 week
  NASA Task Load Index will be queried during a memory task. It includes self-report scales that provide state markers of cognitive effort.
Change in "Time to complete unsolvable anagrams" from baseline | 1 week
  Time in seconds participants spend on unsolvable anagram task before quitting.

SECONDARY OUTCOMES:
Change in "Memory recognition discriminability (d')" from baseline | 1 week
  A standard measure of memory recognition performance in an associative memory task.
Change in "Intrinsic functional connectivity strength" from baseline | 1 week
  A measure of the strength with which mid-cingulate cortex and other brain regions are functionally connected, as measured with resting-state fMRI.
Change in "California Verbal Learning Test" score from baseline | 1 week
  California Verbal Learning Test (CVLT-II) is a comprehensive, detailed assessment of verbal learning and memory deficits in older adolescents and adults. The task asks participants to remember a list of 16 words. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sumientra M Rampersad, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified connectivity maps and motivation and memory task data will be made available via our lab website.
Time Frame: Data will be made available within 6 months after publication.
Access Criteria: Data will be freely available on our lab website.